CLINICAL TRIAL: NCT06990412
Title: A Prospective, Multi-Center Clinical Trial to Evaluate the Safety and Efficacy of an Implantable Wireless Brain-Computer Interface（BCI）System NEO in Patients With Tetraplegia
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of an Implantable Wireless Brain-Computer Interface（BCI）System NEO in Patients With Tetraplegia
Acronym: NEO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuracle Medical Technology(Shanghai) Co.,Ltd. (Industry)
Collaborators: Huashan Hospital (Other); Xuanwu Hospital, Beijing (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Beijing Tiantan Hospital (Other); Henan Provincial People's Hospital (Other); West China Hospital (Other); Affiliated Hospital of Nantong University (Other); The General Hospital of Eastern Theater Command (Other); Peking University Third Hospital (Other); Xiangya Hospital of Central South University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NEURACLE-NEO-202501
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Tetraplegia; Spinal Cord Injuries (SCI)
Keywords: BCI, NEO, Tetraplegia; Spinal cord injury
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: a Minimally Invasive Wireless Implantable Brain-Computer Interface (BCI) System NEO
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): a Minimally Invasive Wireless Implantable Brain-Computer Interface (BCI) System NEO
  Interventions: Device: NEO

INTERVENTIONS:
Device: NEO — a Minimally Invasive Wireless Implantable Brain-Computer Interface (BCI) System NEO

SUMMARY:
To evaluate the safety and efficacy of a Minimally Invasive Wireless Implantable Brain-Computer Interface (BCI) System NEO in patients with tetraplegia and to provide a basis for product registration.

Through brain-computer interface alternative technology, patients can control the external equipment with brain signals to improve the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old, no restriction on gender.
2. Tetraplegia caused by cervical spinal cord injury.
3. Score of ≤1 on either the ball grasp or water pouring tasks of the ARAT (Action Research Arm Test).
4. Muscle strength of finger flexors < grade 3 according to ISNCSCI (International Standards for Neurological Classification of Spinal Cord Injury).
5. Score of ≥2 for "hand to mouth" on ARAT; scores of ≥1 for both "hand to top of head" and "hand to behind the head."
6. Neurological assessment indicates normal function of the motor-related cortex, with no significant structural lesions or functional disorders identified.
7. Diagnosis confirmed for at least 12 months, with a stable condition for at least 6 months following standard treatment.
8. Normal cognitive function, good compliance, and voluntarily agrees to participate in the clinical trial.

Exclusion Criteria:

1. Without the consent of the patient or the patient's legal guardian.
2. Presence of syringomyelia, severe neuropathic pain, or severe spasticity that limits the participant's ability to engage in training.
3. Requires ventilator support.
4. Baclofen dosage >30 mg/day.
5. Received botulinum toxin injections in the upper limb, neck, or hand within 6 months prior to enrollment, or received stem cell therapy within 1 year.
6. High risk of surgical complications, such as active systemic infection, coagulation disorders (e.g., receiving anticoagulant therapy), or platelet count below 50,000.
7. Patients who have already been implanted with medical devices that deliver electrical energy to the central nervous system.
8. Any unstable or significant medical condition that may interfere with study procedures or confound the evaluation of study endpoints, such as depression, mood disorders, or other cognitive impairments.
9. Diagnosed with severe, unstable, and uncontrolled complex regional pain syndrome.
10. Autoimmune-mediated spinal cord dysfunction/injury.
11. History of other neurological disorders, such as stroke, multiple sclerosis, traumatic brain injury, or drug-resistant epilepsy.
12. Peripheral neuropathies (e.g. diabetic polyneuropathy, compressive neuropathies).
13. In the investigator's opinion, the study is unsafe or inappropriate for the participant, or the participant is unlikely to comply with the study follow-up schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
BCI-assisted ARAT grasp response rate | 3 months post-operation
  At 3 months post-operation, the investigator will assess and record the subject's ARAT (Action Research Arm Test) score under BCI-assisted conditions, then compare it with the subject's baseline unassisted ARAT grasp score. The response rate will be calculated as the percentage of responders relative to the total number of participants.
Adverse Events | Immediately post-implantation, and at 3-, and 6-months post-operation.

SECONDARY OUTCOMES:
ISNCSCI Score of the Participant | Baseline, and at 3-, and 6-months post-operation.
  The investigator completes the ISNCSCI (International Standards for Neurological Classification of Spinal Cord Injury) form.
ARAT Score for BCI-Assisted Grasping | 2-, and 6-months post-operation
  The investigator completes the ARAT (Action Research Arm Test) scoring form.
ARAT Score | Baseline, and at 3-, and 6-months post-operation (assessed with the device powered off).
  Investigators will complete the ARAT (Action Research Arm Test) Assessment Form.
Investigator's Overall Device Performance Evaluation | Immediately post-implantation, and at 2-, and 3-, and 6-months post-operation.
  Investigators will complete the Investigator's Overall Device Performance Evaluation Form.
Subject's Overall Device Performance Evaluation | 2-, 3-, and 6-months post-operation.
  Subjects will complete the Subject Device Performance Evaluation Questionnaire.
Device Impedance | 1, 2-, 3-, and 6-months post-operation.
  Record the impedance of each channel; impedance is considered normal if it does not exceed 20 kΩ.
Average Monthly Device Usage Time | 2-, 3-, and 6-months post-operation.
  Calculate the total device usage time per month for each participant.
Participant Quality of Life Score | Baseline, and at 2-, 3-, and 6-months post-operation.
  Assessment Method: Participants complete the "Quality of Life Questionnaire"
Subject Satisfaction Rating | 2-, 3-, and 6-months post-operation.
  Participants evaluate the device's connectivity, operational performance, structural design, and functional design at each follow-up visit.
Investigator Satisfaction with Device Operation | 1-, 2-, 3-, and 6-months post-operation.
  At the 1, 2, 3 and 6-month follow-up visits, investigators evaluate the device's connectivity and stability, as well as its electromagnetic compatibility.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No